CLINICAL TRIAL: NCT05249985
Title: Effects of Protein Supplementation and Neuromuscular Electrical Stimulation on Fat-free Mass in Persons With Motor Complete Spinal Cord Injury: a Pilot Study
Brief Title: Protein Supplementation and Neuromuscular Electrical Stimulation in Persons With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: McMaster University (Other); Danone Nutricia (Industry)
Responsible Party: Principal Investigator, Professor Victoria Tolfrey, Professor of Applied Disability Sport Director of the Peter Harrison Centre for Disability Sport, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3176
Record Dates: First submitted 2022-01-27; First posted 2022-02-22 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injuries
Keywords: Protein; NMES
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study. This will be either (a) NMES plus protein supplementation, or (b) NMES only.
Masking Description: As no placebo supplement is being used in this intervention, it is not possible to do any form of masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES plus protein supplementation (Experimental): Participants will undergo 12 weeks of neuromuscular electrical stimulation- (NMES) based resistance training on the quadriceps in addition to a daily protein supplement.
  Interventions: Device: NMES; Dietary Supplement: Protein
- NMES (Active Comparator): Participants will undergo 12 weeks of neuromuscular electrical stimulation- (NMES) based resistance training on the quadriceps.
  Interventions: Device: NMES

INTERVENTIONS:
Device: NMES — Participants will undergo 12 weeks of neuromuscular electrical stimulation- (NMES) based resistance training on the quadriceps.
Dietary Supplement: Protein — Participants will consume a daily protein supplement
  Arms: NMES plus protein supplementation

SUMMARY:
The aim of this pilot study is to explore how body composition, circulating markers of metabolic health and skin integrity in persons with a spinal cord injury (SCI) are affected by 12 weeks of quadriceps neuromuscular electrical stimulation (NMES) resistance training. The novel element of this study is that one group will be given additional daily protein supplementation in addition to the NMES training (treatment group), whereas the other group will only perform the NMES training (control group). The investigators hypothesise that NMES in combination with protein results in larger improvements in the aforementioned outcomes compared with NMES alone.

DETAILED DESCRIPTION:
A spinal cord injury (SCI) is a debilitating condition, with paralysis below the lesion level as one of the main hallmarks. As a result of paralysis, together with decreased levels of physical activity and impairment-specific co-morbidities such as autonomic dysfunction, persons with SCI have a markedly reduced muscle mass. Being the major site for glucose disposal, skeletal muscle is key for the maintenance of metabolic health, while it also helps with weight management by contributing to energy expenditure at rest. As such, effective strategies to restore muscle mass in persons with SCI are warranted and can have a significant impact on metabolic health and chronic disease risk in this population.

While resistance training is widely recognised as an effective intervention to increase muscle mass in able-bodied individuals, paralysis in the lower limbs of persons with SCI precludes the use of traditional resistance training in this population. NMES has been developed to overcome this barrier and allows persons with SCI to engage in resistance exercise. Notwithstanding the evidence supporting the use of NMES on its own, combined interventions may further enhance its potential to improve health and physical function. Indeed, in the more widely studied population of older adults, that is also at risk for sarcopenia (loss of skeletal muscle mass and strength), increasing daily protein intake enhances the efficacy of resistance training to increase muscle mass.

The primary objective of this study is to determine the impact of a 12-week intervention of NMES in combination with protein supplementation when compared with NMES alone on fat free mass in the legs. Secondary objectives are to investigate the impact of the intervention on 1) markers of cardiometabolic health, namely glucose tolerance and fasting plasma lipid concentrations, 2) resting metabolic rate, and 3) skin blood flow at the level of the sacrum in response to experimental pressure. Outcomes related to tertiary objectives include perceived quality of life, neuropathic pain, body image, sleep quality and spasms; as well as free-living energy balance, physical activity and feasibility outcomes related to recruitment, adherence and participant' experiences with the intervention. It is hypothesised that NMES in combination with protein results in larger improvements in the aforementioned outcomes compared with NMES alone.

ELIGIBILITY:
Inclusion Criteria:

* Motor complete spinal cord injury
* Time since injury injury >1 year

Exclusion Criteria:

* Spinal cord injury below T10 vertebrae
* Habitual protein intake exceeding 2g / kg body mass / day
* Having used NMES resistance training once or more per week in the last six months
* Lactose intolerant
* Any disease or medication that means the participant should not exercise
* Participation in a study involving ionising radiation in the previous 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Dual x-ray absorptiometry
Change in lean soft tissue mass | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Dual x-ray absorptiometry
Change in fat mass | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Dual x-ray absorptiometry

SECONDARY OUTCOMES:
Change in glucose tolerance | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Oral glucose tolerance test
Change in insulin resistance | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Oral glucose tolerance test
Change in fasting plasma lipid concentrations | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Resting blood sample
Change in fasting circulating C-reactive protein | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Resting blood sample
Change in sacral skin blood flow | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Doppler flowmetry
Change in resting metabolic rate | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Expired air analysis

OTHER OUTCOMES:
Change in blood pressure | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Automatic blood pressure cuff
Change in daily energy intake | Pre-intervention (baseline) and at 1 week post-12 week intervention
  3 day food diary
Change in physical activity | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Wrist-worn accelerometer
Change in physical activity | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Leisure time physical activity questionnaire
Change in sleep efficiency and duration | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Wrist-worn accelerometer
Change in sleep quality | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Sleep Quality Scale (available answers include: rarely, sometimes, often, almost always)
Change in muscle spasticity | Pre-intervention (baseline) and at 1 week post-12 week intervention
  The Spinal Cord Injury Spasticity Evaluation Tool
Change in mental health | Pre-intervention (baseline) and at 1 week post-12 week intervention
  5-item Mental Health Inventory
Change in neuropathic pain | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Neuropathic Pain Questionnaire
Change in body image | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Body Image Satisfaction Questionnaire
Change in skinfold thickness | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Measured in millimetre
Height | Pre-intervention only
  Measured in meters
Change in waist and hip circumference | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Measured in centimeters to provide a waist-to-hip ratio
Change in body weight | Pre-intervention (baseline) and at 1 week post-12 week intervention
  Measured in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom